CLINICAL TRIAL: NCT05253664
Title: Evaluation of the Effect of Woman-Centered Care Given in the Early Postpartum Period on Anxiety and Comfort Levels
Brief Title: Effect of Woman-Centered Care on Anxiety and Comfort Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Woman-Cent. Care on Anx.
Record Dates: First submitted 2022-02-02; First posted 2022-02-24 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2022-02

CONDITIONS: Anxiety State; Condition; Physical Suffering
Keywords: Postpartum; woman-centered care; Standard care; comfort; anxiety
MeSH Terms: conditions — Anxiety Disorders; Disease; Pain

STUDY DESIGN:
Intervention Model Description: The study was conducted as a single blind, prospective, and simple randomized controlled trial. The sample was calculated through Power analysis. In the power analysis, the sample size was calculated as a minimum of 105 for each group, according to α:0.05 and 1-β= 0.95. Considering the possibility of loss or separation of the selected specimens during the conduct of the study, 240 women who met the inclusion criteria were assigned to the experimental (120) and control (120) groups. The size and number of blocks divided into two groups as E and C was calculated as 20 (6E and 6C) with twelve mothers in each block. Using Microsoft Office Excel 2016, numbers ranging from 1 to 20 were randomly generated. A total of 240 mothers were evenly assigned to both groups. At the time of the study, 22 women were excluded from the study. The research was completed with 218 mothers, 109 women in each of the experimental and control groups.
Who Masked: Participant
Masking Description: Participants didn't know which group they were allocated. The participants will be blind when they take Woman-Centered Care from investigators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Woman-Centered Care Group (Experimental): Woman-centered care was given to the experimental group. At the time of the study, 6 women were discharged early, 4 women did not want to continue the study, and the babies of 1 women were admitted to the neonatal intensive care unit due to complications so these women were excluded from the study. The study was completed with 109 women in the experimental group.
  Interventions: Behavioral: Woman-Centered Care Group
- Control Group (No Intervention): Standard care was given to the control group. At the time of the study, 2 women were discharged early, 7 women did not want to continue the study, and the babies of 2 women were admitted to the neonatal intensive care unit due to complications so these women were excluded from the study. The study was completed with 218 mothers, with 109 women in the control group.

INTERVENTIONS:
Behavioral: Woman-Centered Care Group — Each woman in the experimental group was given woman-centered care as from 2 hours postpartum and this process continued until 24 hours postpartum. Physiological parameters (systolic-diastolic blood pressure, pulse, body temperature) of women assigned either to the experimental group or the control group were measured at 2 hrs postpartum. The State, Trait Anxiety, and Postpartum Comfort Scales were pretested. A dynamic interaction was ensured between the researcher and the women in the experimental group who received woman-centered care. In the processes of determining and meeting the care needs of women in the early postpartum period, both the women and the researcher took equal responsibilities and the common goal of achieving safe results was shared. Clinical guidelines were used while providing woman-centered care.
  Arms: Woman-Centered Care Group

SUMMARY:
H1a: There is a statistically significant difference in anxiety levels between women who received woman-centered care in the early postpartum period and women who received standard care.

H1b: There is a statistical difference in terms of comfort levels between women who received woman-centered care in the early postpartum period and women who received standard care.

H0a: There is no statistically significant difference in anxiety levels between women who received woman-centered care in the early postpartum period and women who received standard care.

H0b: There is no statistical difference in terms of comfort levels between women who receive female-centered care in the early postpartum period and women who receive standard care.

DETAILED DESCRIPTION:
The research was carried out as a single-blind and block randomized control. The research was conducted in a tertiary hospital in Turkey between February, 2019 and February 2020. The universe of the research consisted of women who gave birth by cesarean section. In the power analysis, the sample size was calculated as a minimum of 105 for each group, according to α:0.05 and 1-β= 0.95. Considering the possibility of loss or separation of the selected specimens during the conduct of the study, 240 women who met the inclusion criteria were assigned to the experimental (120) and control (120) groups.Due to the nature of the study, it was conducted as a single-blind randomized controlled trial.

The pre-test procedure was performed when the mothers' statuses were stabilized two hour after the admittance to the maternity service. The post-test procedure was conducted one hour before the discharge. Woman-centered care was provided to the experimental group, and standard care was provided to the control group.The women in the experimental and control groups were not told which group they were in. Each woman in the experimental group was given woman-centered care from the 2nd hour postpartum, and this process continued until the mother was discharged (mothers are discharged after 24 hours). The standard care provided by the hospital covers the basic postpartum care components. These components are the nutrition of the newborn and the protection of maternal and newborn health. A dynamic interaction was established between the women in the experimental group and the researcher in which woman-centered care was applied. Each woman in the experimental group was responsible for explaining herself, her own health behaviors, and her own needs and values.

"Descriptive Information Form", "Postpartum Comfort Scale" and "State-Trait Anxiety Inventory" were used as data collection tools.

Statistical analyses were performed using IBM SPSS (Statistical Package for Social Sciences) Statistics 22 software. Descriptive statistics (mean, standard deviation, frequency and percentage values) were used to assess the results. Kolmogorov-Smirnov test was used to review the goodness of fit to normal distribution.

ELIGIBILITY:
Inclusion Criteria:

* To receive woman-centered care
* To have cesarian section
* To have singleton birth
* To be within the early postpartum period (the first 24 hours)
* Not have complications childbirth
* Not have chronic diseases or mental disorders
* Older than 18 years
* To voluntary to participate
* To know how to read, write and speak in Turkish
* To stay within this study until the end
* To fully complete questionnaire
* To have a newborn with no complications
* To have a healthy baby

Exclusion Criteria:

* To receive standart care
* Not have cesarian section
* Having multiple birth
* Not to be within the early postpartum period (the first 24 hours)
* Having complications childbirth
* Having chronic diseases or mental disorders
* Younger than 18 years
* To refuse to participate
* Not knowing how to read, write and speak Turkish
* To leave early this study
* Not fill the questionnaire
* Having a newborn with complications
* Having a baby in need of medical care

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2020-02-11 (Actual)

PRIMARY OUTCOMES:
Pre-Test State, Trait Anxiety | 2nd postpartum hour
  The State, Trait Anxiety Inventory consists of two subscales, being state and trait anxiety subscales, and 40 items. The State Anxiety Inventory determines how an individual feels at a certain moment and under certain conditions, and the Trait Anxiety Inventory on the other hand, generally determines how one feels. High scores indicate a high level of anxiety.
Postpartum Comfort Scale | 2nd postpartum hour
  It is a five-point Likert-type scale that evaluates the physical, psychological, sociocultural and environmental comfort of mothers who had cesarean section and normal spontaneous delivery. The lowest and the highest scores that can be obtained from the 34-item scale are 34 and 170, respectively. High scores obtained from the scale indicate that the level of comfort increases.
Systolic blood pressure | 2nd postpartum hour
  All of women were measured from the cubital fossa area using a digital sphygmomanometer. In order to ensure consistency in the measurement of physiological parameters, measurements were conducted on the women using the same devices. The first measurement of the physiological parameters of the women in both the experimental and control groups was recorded when they agreed to participate in the study. The measurement taken at the 2nd postpartum hour will be accepted. It will not be combined with the value measured at another time.
Diastolic blood pressure | 2nd postpartum hour
  All of women were measured from the cubital fossa area using a digital sphygmomanometer. In order to ensure consistency in the measurement of physiological parameters, measurements were conducted on the women using the same devices. The first measurement of the physiological parameters of the women in both the experimental and control groups was recorded when they agreed to participate in the study. The measurement taken at the 2nd postpartum hour will be accepted. It will not be combined with the value measured at another time.
Pulse | 2nd postpartum hour
  Pulse was measured using a digital sphygmomanometer. In order to ensure consistency in the measurement of physiological parameters, measurements were conducted on the women using the same devices. The first measurement of the physiological parameters of the women in both the experimental and control groups was recorded when they agreed to participate in the study. The measurement taken at the 2nd postpartum hour will be accepted. It will not be combined with the value measured at another time.
Body temperature | 2nd postpartum hour
  Body temperature was measured from the forehead using a non-contact thermometer. In order to ensure consistency in the measurement of physiological parameters, measurements were conducted on the women using the same devices. The first measurement of the physiological parameters of the women in both the experimental and control groups was recorded when they agreed to participate in the study. The measurement taken at the 2nd postpartum hour will be accepted. It will not be combined with the value measured at another time.

SECONDARY OUTCOMES:
Post-Test State, Trait Anxiety | 24th postpartum hour
  The State, Trait Anxiety Inventory consists of two subscales, being state and trait anxiety subscales, and 40 items. The State Anxiety Inventory determines how an individual feels at a certain moment and under certain conditions, and the Trait Anxiety Inventory on the other hand, generally determines how one feels. High scores indicate a high level of anxiety.
Post-Test postpartum Comfort Scale | 24th postpartum hour
  It is a five-point Likert-type scale that evaluates the physical, psychological, sociocultural and environmental comfort of mothers who had cesarean section and normal spontaneous delivery. The lowest and the highest scores that can be obtained from the 34-item scale are 34 and 170, respectively. High scores obtained from the scale indicate that the level of comfort increases.
Systolic blood pressure | 20th postpartum hour
  All of women were measured from the cubital fossa area using a digital sphygmomanometer. In order to ensure consistency in the measurement of physiological parameters, measurements were conducted on the women using the same devices. The measurement taken at the 20th postpartum hour will be accepted. It will not be combined with the value measured at another time.
Diastolic blood pressure | 20th postpartum hour
  All of women were measured from the cubital fossa area using a digital sphygmomanometer. In order to ensure consistency in the measurement of physiological parameters, measurements were conducted on the women using the same devices. The measurement taken at the 20th postpartum hour will be accepted. It will not be combined with the value measured at another time.
Pulse | 20th postpartum hour
  Pulse was measured using a digital sphygmomanometer. In order to ensure consistency in the measurement of physiological parameters, measurements were conducted on the women using the same devices. The measurement taken at the 20th postpartum hour will be accepted. It will not be combined with the value measured at another time.
Body temperature | 20th postpartum hour
  Body temperature was measured from the forehead using a non-contact thermometer. In order to ensure consistency in the measurement of physiological parameters, measurements were conducted on the women using the same devices. The measurement taken at the 20th postpartum hour will be accepted. It will not be combined with the value measured at another time.

CONTACTS AND LOCATIONS:
Overall Officials: Aysegul Durmaz, Ph.D., Principal Investigator — Kutahya Health Science University
Locations (1):
- Kutahya Health Science University, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Starting 6 months after publication
Access Criteria: If study' IPD are used, my article should be cited.

REFERENCES:
- [Result] Durmaz A, Komurcu N. Relationship Between Maternal Characteristics and Postpartum Hemorrhage: A Meta-Analysis Study. J Nurs Res. 2018 Oct;26(5):362-372. doi: 10.1097/jnr.0000000000000245. PMID 29219937
- [Result] Finlayson K, Crossland N, Bonet M, Downe S. What matters to women in the postnatal period: A meta-synthesis of qualitative studies. PLoS One. 2020 Apr 22;15(4):e0231415. doi: 10.1371/journal.pone.0231415. eCollection 2020. PMID 32320424
- [Result] Ceylan B, Eser I. Assessment of individualized nursing care in hospitalized patients in a university hospital in Turkey. J Nurs Manag. 2016 Oct;24(7):954-961. doi: 10.1111/jonm.12400. Epub 2016 Jun 14. PMID 27297976
- [Result] Verbiest S, Tully K, Simpson M, Stuebe A. Elevating mothers' voices: recommendations for improved patient-centered postpartum. J Behav Med. 2018 Oct;41(5):577-590. doi: 10.1007/s10865-018-9961-4. Epub 2018 Aug 9. PMID 30094530
- [Result] Fontein-Kuipers Y, de Groot R, van Staa A. Woman-centered care 2.0: Bringing the concept into focus. Eur J Midwifery. 2018 May 30;2:5. doi: 10.18332/ejm/91492. eCollection 2018. PMID 33537566
- [Result] Verbiest S, Bonzon E, Handler A. Postpartum Health and Wellness: A Call for Quality Woman-Centered Care. Matern Child Health J. 2016 Nov;20(Suppl 1):1-7. doi: 10.1007/s10995-016-2188-5. PMID 27757754